CLINICAL TRIAL: NCT06643442
Title: Repurposing Empagliflozin for Duchenne Muscular Dystrophy - Associated Cardiomyopathy: a Pharmacokinetics, Safety and Proof-of-concept Study Among Children 6-18 Years of Age
Brief Title: Repurposing Empagliflozin for DMD-associated Cardiomyopathy in Children 6-18 Years of Age
Acronym: REDMeD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sebastiano Lava (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University College, London (Other); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor-Investigator, Sebastiano Lava, Chief Investigator, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24HL14; 2024-000201-33 (EudraCT Number)
Record Dates: First submitted 2024-06-03; First posted 2024-10-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-10

CONDITIONS: DMD-associated Dilated Cardiomyopathy
MeSH Terms: conditions — Dmd-Associated Dilated Cardiomyopathy | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin (Experimental): All participants will receive the IMP (open-label trial, primary outcome PK)
  Interventions: Drug: Empagliflozin Tablets

INTERVENTIONS:
Drug: Empagliflozin Tablets — Empagliflozin 10mg p.o. once daily (commercially available tablet)

SUMMARY:
This study aims at exploring the use of empagliflozin in children and adolescents 6-18 years old with Duchenne muscular distrophy (DMD) - associated cardiomyopathy. This molecule is effective in reducing hospitalizations and mortality in adults with heart failure and is used in adolescents with type 2 diabetes mellitus, but little is known on children and adolescents with heart failure. Particularly, the best dose to use in this population is currently unknown. This trial aims to:

1. define a dose rationale for this indication and age group (pharmacokinetic study),
2. assess and monitor safety,
3. assess ease-of-swallow,
4. explore middle-term (3-6 months) efficacy and efficacy markers.

Participants will be asked to attend 5 study visits over 6 months, and one end-study visit 2-12 weeks thereafter. Visit 1 will entail an 8h day-hospital stay, while Visits 2, 3, 4 and 5, as well as the end-study visit, will be outpatient clinics (approximately 2h). Participants will be asked to take the studied drug once daily during the 6 months of the study period.

No comparison group is foreseen for this study.

DETAILED DESCRIPTION:
Cardiac disease represents the main life-limiting condition in Duchenne muscular dystrophy (DMD). It is important to recognize and address this early in the disease course. Because of lack of DMD specific drugs, present attitudes for established DMD-related cardiomyopathy ground on current treatment for heart failure. Unfortunately, however, current heart failure therapy in Paediatrics is still unsatisfactory, with high in-hospital (7-26%), and 5-year mortality (30%-50%). Furthermore, mortality rate for DMD cardiomyopathy is worse than similarly aged idiopathic dilated cardiomyopathy (DCM) patients.

Among the recent improvements in adult heart failure management, the sodium glucose transporter type 2 inhibitors (SGLT2i) dapagliflozin and empagliflozin were found to reduce cardiovascular death or worsening heart failure by 25% on top of optimal medical therapy. Indeed, since 2021, they have been recommended as part of standard heart failure therapy.

In the past, paediatric heart failure trials often failed, mainly because of suboptimal dose or inappropriate formulations and endpoints.

This phase II.a, open-label trial is designed to characterize pharmacokinetics (primary outcome), ease-of-swallow, safety and explore potential efficacy markers (secondary outcomes) of empagliflozin in 12 children and adolescents with DMD-related cardiomyopathy, so to inform the design and performance of subsequent, state-of-the-art, high-quality efficacy trials.

Participants will receive empagliflozin during 6 months. They will have 5 visits, one end-study visit and 7 to 8 pharmacokinetic samples. The timing of these samples will be optimized exploiting contemporary modeling and simulation techniques.

Safety evaluation will occur throughout the study, while ease-of-swallow will be evaluated at Visit 1, and efficacy markers at Visits 1, 4 and 5.

Pharmacokinetic modeling will characterize primary and secondary pharmacokinetic parameters and allow to define the optimal paediatric dose, informing both current compassionate-care use and the design of future efficacy trials.

ELIGIBILITY:
Inclusion Criteria:

* Children or adolescents 6 to 18 years of age with DMD-associated cardiomyopathy, followed either as in- or outpatients, will be eligible for inclusion.
* Currently on heart failure medication (any drug or any combination).
* Patients should potentially benefit from adding a SGLT2i (as judged by the treating physician and the PI or Co-PI).
* Patients need to be on stable medical treatment, defined as no new heart failure drug started over the preceding 2 weeks and no major drug dose modification (apart minor adaptations, like weight adaptations, rounding or formulation changes) during the 2 weeks prior to enrolment.
* Adolescents, respectively parents or caregivers of children, capable of giving informed consent.
* Ability to tolerate a cardiac MRI investigation without the need of general anaesthesia.

Exclusion Criteria:

* Inability to understand and go through the informed consent procedure.
* Inability to receive medications per os or through a nasogastric tube.
* Type 1 or Type 2 Diabetes mellitus or any underlying metabolic disease associated with hypoglycaemias.
* Body weight <15kg.
* Current smokers (defined as >1 cigarette/week).
* Use of any other nicotine-delivering product (e.g. nicotine patches).
* Any known illicit drug abuse.
* Active chronic HBV, HCV or HIV.
* Any major surgery within 4 weeks of first dose administration.
* Blood transfusion recipient within 4 weeks of dose administration.
* eGFR <45mL/min/1.73m2 (simplified Schwartz formula or Filler formula).
* K+ >6.5mmol/L.
* Blood glucose <4mmol/L.
* There are no blood pressure exclusion criteria foreseen, but participants need to be haemodynamically stable, as assessed by the local investigator.
* Sustained or symptomatic arrhythmia insufficiently controlled with drug and/or device therapy.
* Cardio-surgical procedure within the 2 months prior to Visit 1, or interventional cardiac catheterization within 2 weeks prior to Visit 1, or the patient is planned to undergo cardiac surgery or an interventional cardiac catheterization during the study period (i.e. in the 6 months following Visit 1).
* Post-menarchal female patients of childbearing potential cannot be included. Participants who begin menstruating during the trial will be discontinued from the IMP. However, their monitoring will continue up to 6 months after their first dose of IMP.
* Known lactose intolerance, galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption.
* Known allergies to active ingredients or excipients of commercially available empagliflozin tablets.
* Significant medical history of active severe medical disease.
* Significant liver disease, Child Pugh Class C, or significant laboratory abnormalities at enrolment.
* Significant gastroenterological or hepatic disease that could significantly impair absorption or metabolism of orally administered drugs.
* Any medical co-morbidity, which is deemed incompatible (or only with relevant risk) with study participation by the treating clinician and/or the study investigator.
* Active urinary tract infection (being treated with antibiotics at the moment of Visit 1) or other relevant bacterial infection, as judged by the treating clinician and/or the study investigator.
* The patient is currently participating in another interventional clinical trial or has participated in such a trial during the <14 days before Visit 1 (or if enrolment in this study is incompatible with the protocol of that preceding trial), or the duration of five half-lives of the IMP, whichever is longer.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics - apparent clearance (CL/F) | Visit 1 to Visit 3 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks after study start)
  Empagliflozin concentrations at the different time-points (6 samples at Visit 1, 1 opportunistic sample at Visits 2 and 3; the timing of the samples will be optimized with modeling & simulation techniques).
  Basing on these concentrations, non-compartmental pharmacokinetic calculations will be performed, allowing to determine pharmacokinetic parameters (including CL/F).
Pharmacokinetics - apparent (central) volume of distribution (Vd/F) | Visit 1 to Visit 3 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks after study start)
  Empagliflozin concentrations at the different time-points (6 samples at Visit 1, 1 opportunistic sample at Visits 2 and 3; the timing of the samples will be optimized with modeling & simulation techniques).
  Basing on these concentrations, non-compartmental pharmacokinetic calculations will be performed, allowing to determine pharmacokinetic parameters (including Vd/F).
Pharmacokinetics - half-life | Visit 1 to Visit 3 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks after study start)
  Empagliflozin concentrations at the different time-points (6 samples at Visit 1, 1 opportunistic sample at Visits 2 and 3; the timing of the samples will be optimized with modeling & simulation techniques).
  Basing on these concentrations, non-compartmental pharmacokinetic calculations will be performed, allowing to determine pharmacokinetic parameters (including t1/2).
Pharmacokinetics - AUC | Visit 1 to Visit 3 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks after study start)
  Empagliflozin concentrations at the different time-points (6 samples at Visit 1, 1 opportunistic sample at Visits 2 and 3; the timing of the samples will be optimized with modeling & simulation techniques).
  Basing on these concentrations, non-compartmental pharmacokinetic calculations will be performed, allowing to determine pharmacokinetic parameters (including AUC).
Pharmacokinetics - maximal concentration (Cmax) | Time Frame: Visit 1 to Visit 3 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks after study start)
  Empagliflozin concentrations at the different time-points (6 samples at Visit 1, 1 opportunistic sample at Visits 2 and 3; the timing of the samples will be optimized with modeling & simulation techniques).
  Basing on these concentrations, non-compartmental pharmacokinetic calculations will be performed, allowing to determine pharmacokinetic parameters (including Cmax).

SECONDARY OUTCOMES:
Safety 1 - eGFR | Visit 1 to Visit 5 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months after enrolment)
  Creatinine, respectively Cystatin C, will be collected in order to calculate eGFR (bedside Schwartz formula, respectively Filler equation).
Safety 2 - Occurrence of hypoglycemia | Visit 1 to Visit 5 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months after enrolment)
  Blood glucose will be checked three times at Visit 1 (baseline, at approximately 2-3h post-intake, and before discharge at 8h post-intake), as well as once at Visits 2 to 5. Outcome measure: number of patients experiencing hypoglycemia.
Safety 3 - Occurrence of ketoacidosis | Visit 1 to Visit 5 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months after enrolment)
  The outcome is presence (or absence) of ketoacidosis. This will be assessed at Visits 1, 2, 3, 4 and 5. Outcome measure: number of patients experiencing ketoacidosis.
Safety 4 - Occurrence of UTI | Visit 1 to Visit 5 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months after enrolment)
  The outcome is presence (or absence) of UTI diagnosis. This will be assessed at Visits 1, 2, 3, 4 and 5. Outcome measure: number of patients experiencing UTI between Visit 2 and Visit 5.
Ease of swallow | Visit 1 (Visit 1 = day 1)
  Ease of swallow will be assessed by means of facial hedonic scales, according to our standard procedure, at Visit 1. (Scale 1 to 4, 1 being the worse and 4 the best score: very difficult - difficult - possible - easy to swallow.)
Efficacy and efficacy markers (exploratory) 1 - Heart failure severity class | Visit 1 to Visit 5 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months after enrolment)
  Symptoms, clinical signs, NYHA (if > or =8 years of age) / Ross (if <8 years of age) class assignment. NYHA and Ross heart failure classes share the same scale of I (no limitation of physical activity) to IV (symptoms at rest). Analysis will be performed at Visit 1, Visit 4 and Visit 5. Outcome: change between Visit 1 and Visit 5.
Efficacy and efficacy markers (exploratory) 2 - NT-proBNP level | Visit 1 to Visit 5 (Visit 1 = day 1, Visit 2 = 1 week, Visit 3 = 5-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months after enrolment)
  Analysis will be performed at Visits 1, 3, 4 and 5. Outcome: change between Visit 1 and Visit 5.
Efficacy and efficacy markers (exploratory) 3 - Echocardiography 1: Left-ventricular end-diastolic diameter (LVEDd) | Visits 1, 4 and 5 (Visit 1 = day 1, Visit 4 = 3 months, Visit 5 = 6 months after enrolment)
  LVEDd (z-score) will be measured at Visits 1, 4 and 5. Outcome: change between Visit 1 and Visit 5.
Efficacy and efficacy markers (exploratory) 4 - Echocardiography 2: Left-ventricular end-systolic diameter (LVESd) | Visits 1, 4 and 5 (Visit 1 = day 1, Visit 4 = 3 months, Visit 5 = 6 months after enrolment)
  LVESd (z-score) will be measured at Visits 1, 4 and 5. Outcome: change between Visit 1 and Visit 5.
Efficacy and efficacy markers (exploratory) 5 - Echocardiography 3: Fractional shortening (FS) | Visits 1, 4 and 5 (Visit 1 = day 1, Visit 4 = 3 months, Visit 5 = 6 months after enrolment)
  FS (%) will be measured at Visits 1, 4 and 5. Outcome: change between Visit 1 and Visit 5.
Efficacy and efficacy markers (exploratory) 6 - Echocardiography 4: Left ventricular ejection fraction (LV-EF) | Visits 1, 4 and 5 (Visit 1 = day 1, Visit 4 = 3 months, Visit 5 = 6 months after enrolment)
  LV-EF (%) will be measured at Visits 1, 4 and 5. Outcome: change between Visit 1 and Visit 5.
Efficacy and efficacy markers (exploratory) 7 - cMRI 1: Left ventricular end-diastolic volume | Visit 1, Visit 5 (Visit 1 = day 1, Visit 5 = 6 months after enrolment)
  LV end-diastolic volume will be measured at Visits 1 and 5. Outcome: change between Visit 1 and Visit 5.
Efficacy and efficacy markers (exploratory) 8 - cMRI 2: Left ventricular end-systolic volume | Visit 1, Visit 5 (Visit 1 = day 1, Visit 5 = 6 months after enrolment)
  LV end-systolic volume will be measured at Visits 1 and 5. Outcome: change between Visit 1 and Visit 5.
Efficacy and efficacy markers (exploratory) 9 - cMRI 3: Left ventricular ejection fraction | Visit 1, Visit 5 (Visit 1 = day 1, Visit 5 = 6 months after enrolment
  LV end-systolic ejection fraction will be measured/calculated at Visits 1 and 5. Outcome: change between Visit 1 and Visit 5.
Efficacy and efficacy markers (exploratory) 10 - cMRI 4: Presence of late gadolinium enhancement | Visit 1, Visit 5 (Visit 1 = day 1, Visit 5 = 6 months after enrolment)
  Presence (y) or absence (n) of late gadolinium enhancement in each of the 17 AHA segments will be measured at Visits 1 and 5. Outcome: change in number of LGE positive segments between Visit 1 and Visit 5.
Efficacy and efficacy markers (exploratory) 11 - cMRI 5: Extracellular volume (ECV) | Visit 1, Visit 5 (Visit 1 = day 1, Visit 5 = 6 months after enrolment)
  Extracellular volume (ECV) will be measured/calculated at Visits 1 and 5. Outcome: change between Visit 1 and Visit 5.

OTHER OUTCOMES:
Efficacy markers (exploratory), Mechanistic insights - 1: body weight (kg) | Visit 1 to Visit 5 (Visit 2 = 1 week, Visit 3 = 4-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months)
  To explore the effect of SGLT2 inhibitors on fluid status, body weight will be assessed (outcome: change between Visit 1 and Visit 5).
Efficacy markers (exploratory), Mechanistic insights - 2: heart rate (bpm) | Visit 1 to Visit 5 (Visit 2 = 1 week, Visit 3 = 4-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months)
  To explore the effect of SGLT2 inhibitors on sympathetic activation, heart rate (in bpm) will be assessed (outcome: change between Visit 1 and Visit 5).
Efficacy markers (exploratory), Mechanistic insights - 3: blood pressure (SBP/DBP, mmHg) | Visit 1 to Visit 5 (Visit 2 = 1 week, Visit 3 = 4-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months)
  To explore the effect of SGLT2 inhibitors on sympathetic activation, blood pressure (SBP and DBP, in mmHg) will be assessed (outcome: change between Visit 1 and Visit 5).
Efficacy markers (exploratory), Mechanistic insights - 4: b-hydroxybutyrate (mmol/L) | Visit 1 to Visit 5 (Visit 2 = 1 week, Visit 3 = 4-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months)
  To explore the effect of SGLT2 inhibitors on metabolism shift, b-hydroxybutyrate will be assessed (outcome: change between Visit 1 and Visit 5).
Efficacy markers (exploratory), Mechanistic insights - 5: haemoglobin (g/L) | Visit 1 to Visit 5 (Visit 2 = 1 week, Visit 3 = 4-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months)
  To explore the effect of SGLT2 inhibitors on haemoglobin, haemoglobin will be assessed (outcome: change between Visit 1 and Visit 5).
Efficacy markers (exploratory), Mechanistic insights - 6: uric acid (mmol/L) | Visit 1 to Visit 5 (Visit 2 = 1 week, Visit 3 = 4-6 weeks, Visit 4 = 3 months, Visit 5 = 6 months)
  To explore the effect of SGLT2 inhibitors on uric acid homeostasis, uric acid will be assessed (outcome: change between Visit 1 and Visit 5).

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital NHS Foundation Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adorisio R, Mencarelli E, Cantarutti N, Calvieri C, Amato L, Cicenia M, Silvetti M, D'Amico A, Grandinetti M, Drago F, Amodeo A. Duchenne Dilated Cardiomyopathy: Cardiac Management from Prevention to Advanced Cardiovascular Therapies. J Clin Med. 2020 Oct 1;9(10):3186. doi: 10.3390/jcm9103186. PMID 33019553
- [Background] Das BB. Current State of Pediatric Heart Failure. Children (Basel). 2018 Jun 28;5(7):88. doi: 10.3390/children5070088. PMID 29958420
- [Background] Rossano JW, Kim JJ, Decker JA, Price JF, Zafar F, Graves DE, Morales DL, Heinle JS, Bozkurt B, Towbin JA, Denfield SW, Dreyer WJ, Jefferies JL. Prevalence, morbidity, and mortality of heart failure-related hospitalizations in children in the United States: a population-based study. J Card Fail. 2012 Jun;18(6):459-70. doi: 10.1016/j.cardfail.2012.03.001. Epub 2012 Apr 10. PMID 22633303
- [Background] Andrews RE, Fenton MJ, Dominguez T, Burch M; British Congenital Cardiac Association. Heart failure from heart muscle disease in childhood: a 5-10 year follow-up study in the UK and Ireland. ESC Heart Fail. 2016 Jun;3(2):107-114. doi: 10.1002/ehf2.12082. Epub 2016 Jan 24. PMID 27812385
- [Background] Towbin JA, Lowe AM, Colan SD, Sleeper LA, Orav EJ, Clunie S, Messere J, Cox GF, Lurie PR, Hsu D, Canter C, Wilkinson JD, Lipshultz SE. Incidence, causes, and outcomes of dilated cardiomyopathy in children. JAMA. 2006 Oct 18;296(15):1867-76. doi: 10.1001/jama.296.15.1867. PMID 17047217
- [Background] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Background] Bourke JP, Bueser T, Quinlivan R. Interventions for preventing and treating cardiac complications in Duchenne and Becker muscular dystrophy and X-linked dilated cardiomyopathy. Cochrane Database Syst Rev. 2018 Oct 16;10(10):CD009068. doi: 10.1002/14651858.CD009068.pub3. PMID 30326162
- [Background] Muntoni F. Cardiomyopathy in muscular dystrophies. Curr Opin Neurol. 2003 Oct;16(5):577-83. doi: 10.1097/01.wco.0000093100.34793.81. PMID 14501841
- [Background] Bourke J, Turner C, Bradlow W, Chikermane A, Coats C, Fenton M, Ilina M, Johnson A, Kapetanakis S, Kuhwald L, Morley-Davies A, Quinlivan R, Savvatis K, Schiava M, Yousef Z, Guglieri M. Cardiac care of children with dystrophinopathy and females carrying DMD-gene variations. Open Heart. 2022 Oct;9(2):e001977. doi: 10.1136/openhrt-2022-001977. PMID 36252992
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827
- [Background] Braunwald E. Gliflozins in the Management of Cardiovascular Disease. N Engl J Med. 2022 May 26;386(21):2024-2034. doi: 10.1056/NEJMra2115011. No abstract available. PMID 35613023
- [Background] Lava SAG, Laurence C, Di Deo A, Sekarski N, Burch M, Della Pasqua O. Dapagliflozin and Empagliflozin in Paediatric Indications: A Systematic Review. Paediatr Drugs. 2024 May;26(3):229-243. doi: 10.1007/s40272-024-00623-z. Epub 2024 Apr 18. PMID 38635113
- [Background] Verhaert D, Richards K, Rafael-Fortney JA, Raman SV. Cardiac involvement in patients with muscular dystrophies: magnetic resonance imaging phenotype and genotypic considerations. Circ Cardiovasc Imaging. 2011 Jan;4(1):67-76. doi: 10.1161/CIRCIMAGING.110.960740. No abstract available. PMID 21245364
- [Background] Bellanti F, Della Pasqua O. Modelling and simulation as research tools in paediatric drug development. Eur J Clin Pharmacol. 2011 May;67 Suppl 1(Suppl 1):75-86. doi: 10.1007/s00228-010-0974-3. Epub 2011 Jan 19. PMID 21246352
- [Background] Bellanti F, Di Iorio VL, Danhof M, Della Pasqua O. Sampling Optimization in Pharmacokinetic Bridging Studies: Example of the Use of Deferiprone in Children With beta-Thalassemia. J Clin Pharmacol. 2016 Sep;56(9):1094-103. doi: 10.1002/jcph.708. Epub 2016 Apr 1. PMID 26785826
- [Background] Loss KL, Shaddy RE, Kantor PF. Recent and Upcoming Drug Therapies for Pediatric Heart Failure. Front Pediatr. 2021 Nov 11;9:681224. doi: 10.3389/fped.2021.681224. eCollection 2021. PMID 34858897
- [Background] Lava SA, Simonetti GD, Bianchetti AA, Ferrarini A, Bianchetti MG. Prevention of vitamin D insufficiency in Switzerland: a never-ending story. Int J Pharm. 2013 Nov 30;457(1):353-6. doi: 10.1016/j.ijpharm.2013.08.068. No abstract available. PMID 24216246
- [Background] Cella M, Knibbe C, Danhof M, Della Pasqua O. What is the right dose for children? Br J Clin Pharmacol. 2010 Oct;70(4):597-603. doi: 10.1111/j.1365-2125.2009.03591.x. No abstract available. PMID 21087295